CLINICAL TRIAL: NCT07393139
Title: Early Postoperative Pain and Functional Recovery Following a Limb Amputation: a Retrospective Observational Study.
Brief Title: Early Postoperative Pain Following a Limb Amputation
Acronym: Pain-Amp
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 638/2025/Oss/IOR
Record Dates: First submitted 2026-01-16; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Amputation, Surgical; Pain Management; Rehabilitation
Keywords: Phantom limb pain; Amputation; Post-operative
MeSH Terms: conditions — Agnosia; Phantom Limb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amputees: Patients that underwent an amputation to any limb at the IRCCS Istituto Ortopedico Rizzoli between January 1st 2023 and December 31st 2025
  Interventions: Other: Pain assessment

INTERVENTIONS:
Other: Pain assessment — During hospitalization, patients were asked three times daily to rate their pain using the 11 point NRS scale. The highest rating of each day will be extracted from their medical records.

SUMMARY:
The primary aim of this study is to characterize the trajectory of pain and functional recovery in the first post-operative period following a limb amputation. Secondarily, this study aims to conduct an exploratory analysis to evaluate potential associations between clinical, demographical and therapeutical variables and primary outcomes including pain intensity, pain control and functional recovery.

DETAILED DESCRIPTION:
This retrospective observational study will be conducted at IRCCS Istituto Ortopedico Rizzoli. All patients who underwent an amputation at the IRCCS Istituto Ortopedico Rizzoli between January 1st 2023 and December 31st 2025 will be screened for eligibility based on predefined inclusion criteria. Once a patient is included into the study, all relevant data will be collected from their medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Patients who underwent an amputation to any limb, regardless of location or diagnosis

Exclusion Criteria:

* Patients with severe cognitive impairment or diagnosed with dementia
* Patients deceased or in critical conditions within 48 hours of the intervention
* Previous amputation to any limb
* Admission to the hospital because of a stump revision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that underwent an amputation to any limb at the IRCCS Istituto Ortopedico Rizzoli.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | up to 30 days
  Pain intensity was assessed using Numeric Rating Scale (NRS). The NRS is an 11 point scale from 0 to 10, with 0 indicating no pain and 10 representing the worst pain imaginable.

SECONDARY OUTCOMES:
Functional Recovery | up to 30 days
  The number of days required for walking.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Hsu E, Cohen SP. Postamputation pain: epidemiology, mechanisms, and treatment. J Pain Res. 2013;6:121-36. doi: 10.2147/JPR.S32299. Epub 2013 Feb 13. PMID 23426608
- [Background] Kent ML, Hsia HJ, Van de Ven TJ, Buchheit TE. Perioperative Pain Management Strategies for Amputation: A Topical Review. Pain Med. 2017 Mar 1;18(3):504-519. doi: 10.1093/pm/pnw110. PMID 27402960
- [Background] Limakatso K, Ndhlovu F, Usenbo A, Rayamajhi S, Kloppers C, Parker R. The prevalence and risk factors for phantom limb pain: a cross-sectional survey. BMC Neurol. 2024 Feb 6;24(1):57. doi: 10.1186/s12883-024-03547-w. PMID 38321380
- [Background] Moore RA, Chi CC, Wiffen PJ, Derry S, Rice AS. Oral nonsteroidal anti-inflammatory drugs for neuropathic pain. Cochrane Database Syst Rev. 2015 Oct 5;2015(10):CD010902. doi: 10.1002/14651858.CD010902.pub2. PMID 26436601
- [Background] Spezia MC, Dy CJ, Brogan DM. Phantom Limb Pain Management. J Hand Surg Am. 2025 Feb;50(2):208-215. doi: 10.1016/j.jhsa.2024.09.007. Epub 2024 Oct 21. PMID 39436344